CLINICAL TRIAL: NCT06580483
Title: Comparative Assessment of Two Filling Materials As Restorative Options for Tooth-tissue Supported Overdenture: a Split-mouth Randomized Trial
Brief Title: Assessment of Two Filling Materials for Teeth-tissue Supported Overdenture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FODMRC-202100102
Record Dates: First submitted 2024-08-29; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Jaw, Edentulous, Partially
Keywords: overdenture; nanocomposite; Amalgam; Survival; Wear
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A tooth (on one side) supporting complete overdenture (Experimental): The tooth is prepared to receive a restoration
  Interventions: Other: amalgam restoration
- A tooth (on the other side) supporting complete overdenture (Active Comparator): The tooth is prepared to receive another restoration
  Interventions: Other: nano-composite

INTERVENTIONS:
Other: amalgam restoration — An abutment tooth is restored on a side by amalgam plug
  Arms: A tooth (on one side) supporting complete overdenture
Other: nano-composite — An abutment tooth is restored on a side by nano-composite
  Arms: A tooth (on the other side) supporting complete overdenture

SUMMARY:
Methods: 28 patients with bilateral remaining first premolar in the maxillary or mandibular arch were enrolled in the study. Dome shaped preparations of the abutments were performed. The amalgam and composite restorations were randomly assigned to either the right or left remaining premolar; then conventional steps of overdenture fabrication and insertion were accomplished. Patients were followed up for 3 years.

DETAILED DESCRIPTION:
For all cases, root planning and supra- and subgingival scaling were carried out utilizing an ultrasonic scaler. For all cases, all teeth were cleaned, shaped, and obturated during the patients' first visit. Local anaesthesia was achieved by local infiltration. After anaesthesia, an endodontic access cavity was established. Canals were prepared using the crowndown technique. The ideal working length was determined using an electronic apex locator and periapical radiographs. The canals were cleaned and shaped. The final instrumentation size was determined as three sizes larger than the first file binding at the working length. Master apical files ranged from #25 to #50, depending on both root anatomy and initial diameter of the root canal.Irrigation was always performed with 5.25% NaOCl solution. Obturation using gutta-percha. The master gutta-percha cone was coated with AH Plus, obturation was carried out utilizing the lateral compaction technique. Afterwards, selective etching of enamel for 30 seconds then rinsing and dryness were done followed by application of universal bonding agent with agitation action which was then light cured for 20 seconds. It was then followed by core buildup with light cured Nano-filled composite body.. As for the amalgam, high-copper non-gamma 2 spherical and lathe cut amalgam was used. For all patients, fabrication of new dentures was employed.

Data were statistically described in terms of mean, standard deviation (SD), 95% CI, median and range. Data were tested for the normal assumption using Kolmogorov Smirnov test. Comparison between the study groups was done using Student t test for independent samples. Two-sided p values less than 0.05 was considered statistically significant. IBM SPSS. Survival analysis was done using Kaplan Maier statistics

ELIGIBILITY:
Inclusion Criteria:

* Presented with partially edentulous maxillary and mandibular arches particularly with bilaterally remaining any of these teeth ; #33 #34 #35 #43 #44 #45 #13 # 14#15 #23 # 24 #25
* Good periodontal support and grade I mobility.
* They were medically free.

Exclusion Criteria:

* Medically compromised
* Grade II and grade III mobility

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Wear depth | 36 months
  For each patient, a scan of the abutments was performed using intra-oral scanner in the day of overdenture insertion and another scan was performed after 36m follow up periods and then both scans are compared
Survival of the restoration | 36 months
  Restoration survival was assessed according to the criteria approved by the FDI World Dental Federation (FDI) Scientific Committee in 2007 and the General Assembly in 2008 as criteria specifically developed for use in clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Wafaa I Ibrahim, Principal Investigator — Assoc. Prof.
Locations (1):
- Delta University for Science & Technology, Al Mansurah, Egypt